CLINICAL TRIAL: NCT01083212
Title: A Randomised, Open, Placebo Controlled, Two-way Crossover Phase I Study in Type 2 Diabetes Mellitus Patients Treated With Metformin to Evaluate the Effect of Gemfibrozil on the Pharmacokinetics and Pharmacodynamics of a Single Dose of AZD1656
Brief Title: To Evaluate the Effect of Gemfibrozil on the Pharmacokinetics and Pharmacodynamics of a Single Dose of AZD1656
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D1020C00030
Record Dates: First submitted 2010-03-08; First posted 2010-03-09 (Estimated); Last update posted 2010-07-01 (Estimated); Status verified 2010-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Gemfibrozil
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AZD1656; Gemfibrozil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Gemfibrozil day 1-5 + AZD1656 day 4, 1 week without, Placebo day 1-5 + AZD1656 day 4
  Interventions: Drug: AZD1656; Drug: Gemfibrozil; Drug: Placebo
- 2 (Experimental): Placebo day 1-5 + AZD1656 day 4, 1 week without, Gemfibrozil day 1-5 + AZD1656 day 4
  Interventions: Drug: AZD1656; Drug: Gemfibrozil; Drug: Placebo

INTERVENTIONS:
Drug: AZD1656 — Single dose,oral tablet
Drug: Gemfibrozil — Oral tablet bid on day 1 - 5.
Drug: Placebo — Oral tablet bid on day 1-5

SUMMARY:
The purpose of this study is to evaluate the effect of Gemfibrozil on the Pharmacokinetics and Pharmacodynamics of a Single Dose of AZD1656

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed Type 2 diabetes mellitus for at least 1 year and treated with metformin.
* Body mass index between ≥19 and ≤42 kg/m2.

Exclusion Criteria:

* Intake of another investigational drug within the last 30 days prior to enrolment.
* Clinically significant illness or clinically relevant trauma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
PK of AZD1656 when administered with placebo or following repeated dosing of gemfibrozil by assessment of AUC and Cmax. | Serial blood samples will be drawn on day 4-6 period 1 and 2 from pre-dose to 48 h post AZD1656 administration.

SECONDARY OUTCOMES:
PK of AZD1656 when administered with placebo or following repeated dosing of germfibrozil by assessment of AUC0-t, tmax, t1/2, CL/F and Vz/F | Serial blood samples will be drawn on day 4-6 period 1 and 2 from pre-dose to 48 h post AZD1656 administration.
PK of AZD1656 metabolite, when AZD1656 is administered with placebo or following repeated dosing of gemfibrozil by assessment of AUC, AUC0-t, Cmax, tmax, t1/2 | Serial blood samples will be drawn on day 4-6 period 1 and 2 from pre-dose to 48 h post AZD1656 administration.
Safety of AZD1656 when administered with placebo or following repeated dosing of gemfibrozil by assessment of electrocardiogram, weight, pulse, blood pressure, laboratory variables including 24-h plasma glucose, physical examination and adverse events | Paper ECG, BP/pulse preentry, pre-dose,day 4, period 1 and 2, and follow-up on day +7-10 days. Weight, physical examination preentry and pre-dose (period 1 and 2), follow-up. 7-point plasma-glucose on pre-entry, day 3 and 5, period 1 and 2.

CONTACTS AND LOCATIONS:
Overall Officials: Stanko Skrtic, Study Director — AstraZeneca; Aslak Rautio, Principal Investigator — Quintiles Hermelinen AB; Wolfgang Kuhn, Principal Investigator — Quintiles AB; Folke Sjöberg, Principal Investigator — J.J. Berzelius Clinical Research Center AB; Mirjana Kujacic, Study Chair — AstraZeneca
Locations (3):
- Sweden (3):
  - Reserach Site, Linköping
  - Research Site, Luleå
  - Research Site, Uppsala